CLINICAL TRIAL: NCT03591432
Title: A Randomised Controlled Trial Comparing Transnasal humidiﬁed Rapid insufﬂation Ventilatory Exchange (THRIVE) Pre-oxygenation and Apneic Oxygenation With Facemask Pre-oxygenation and Ventilation in Elderly Patients Undergoing Induction of Anaesthesia.
Brief Title: A Trial Comparing Transnasal humidiﬁed Rapid insufﬂation Ventilatory Exchange (THRIVE) and Apneic Oxygenation With Facemask Ventilation in Elderly Patients Undergoing Induction of Anaesthesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Associate Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: THRIVE-ELDERLY
Record Dates: First submitted 2018-07-07; First posted 2018-07-19 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia Intubation Complication; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE (Experimental): Using transnasal humidified rapid insufflation ventilatory exchange (THRIVE) oxygenation technique in elderly patients undergoing induction of anesthesia.
  Interventions: Device: Transnasal humidified rapid insufflation ventilatory exchange (THRIVE)
- Facemask (Active Comparator): Using facemask technique in elderly patients undergoing induction of anesthesia.
  Interventions: Device: Facemask ventilation

INTERVENTIONS:
Device: Transnasal humidified rapid insufflation ventilatory exchange (THRIVE) — Transnasal humidified rapid insufflation ventilatory exchange (THRIVE) is a new technique that is available for use in critically ill patients and in patients with difficult airways. The technique combines the benefits of apneic oxygenation and CPAP with a reduction in CO2 levels through gaseous mixing and flushing of the dead space. THRIVE is administered through a standard, commercially available, nasal, high-flow oxygen delivery system. Insufflation of O2 up to 70 L/min via a purpose-made nasal cannula is used initially to provide preoxygenation, which can be continued during intravenous induction until a definitive airway is secured. The THRIVE technique has been demonstrated to appreciably prolong the safe duration of apnea while avoiding increase in CO2.
  Arms: THRIVE
Device: Facemask ventilation — Nowadays pre-oxygenation is usually achieved using oxygen delivered via a facemask before induction of anaesthesia; this potentially extends the time available for securing the airway before hypoxaemia to 6 min. In patients undergoing elective surgery, the lungs are normally ventilated with a bag/facemask technique after induction, and this can be repeated if attempts at intubating the trachea are prolonged.
  Arms: Facemask

SUMMARY:
Induction of general anaesthesia in patients undergoing emergency surgery can be challenging, because of the often suboptimal circumstances under which anaesthesia has to be delivered, as well as potential physiological derangements caused by their underlying illness, especially in elderly patients. Pre-oxygenation is usually achieved using oxygen delivered via a facemask before induction of anaesthesia. In patients undergoing elective surgery, the lungs are normally ventilated with a bag/facemask technique after induction. However, these options for oxygenation are limited. Facemask ventilation has a perceived risk of gastric insufflation of gas, leading to increased intragastric pressure and raised risk of pulmonary aspiration of stomach contents. Nasal cannulae have been recommended as an alternative method of delivering continuous oxygen during induction of anaesthesia. The Aim of this study is to compare the effect of transnasal humidified rapid insufflation ventilatory exchange (THRIVE) oxygenation with facemask oxygenation on extended apnoeic period and postoperative respiratory complications in elderly patients undergoing induction of anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who required induction of general anaesthesia for emergency surgery, whose routine clinical care required arterial blood gas sampling, and who were competent to give consent were recruited.

Exclusion Criteria:

* Patients who had severe respiratory disease.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative respiratory complications | 14 days after surgery
Extended apnoeic period | during induction of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645